CLINICAL TRIAL: NCT03254251
Title: The Effects of a 12-week Stair Climbing Regimen on Arterial Stiffness, BP and Leg Strength in Stage-1 Hypertensive Postmenopausal Women
Brief Title: The Effects of Stair Climbing on Arterial Stiffness, Blood Pressure and Leg Strength in Stage-1 Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Dong-Eui University (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Won-mok son, postdoctoral fellow, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PusanNU-3
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Hypertension; Menopause
MeSH Terms: conditions — Hypertension | interventions — Stair Climbing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stair Climbing (SC) (Experimental): N=20, 12 weeks of stair climbing exercise training.
  Interventions: Behavioral: Stair climbing
- No Exercise (CON) (No Intervention): N=21, No exercise for 12 weeks

INTERVENTIONS:
Behavioral: Stair climbing — Stair climbing (SC) training was 12 weeks of progressive SC program. Each training session consisted of a general warm-up (5 min: slow and fast skipping, stretching) followed by the SC training and was supervised by experienced personnel. The program began with two bouts of stair climbing four days a week in weeks 1 and 2, increasing by one climb a day every three weeks. By the last three weeks (10-12) of the study, all subjects were completing 5 climbs four days a week. During each climb participants ascended 12 flights (192 steps) divided into 3 sets of 4 flights, with a 2 min rest period between each set. There was a 5 min rest period between climbs that allowed the participants to reach the ground floor using an elevator. Subjects in the non-exercising control group did not participate in a supervised exercise program for the duration of the study.
  Arms: Stair Climbing (SC)

SUMMARY:
We used a parallel experimental design. Following an initial screening and familiarization session of study tests and procedures, eligible postmenopausal women were randomly assigned to a stair climbing (SC) group or non-exercising control group. SC training session was progressive program, and was performed 4 days a week for 12 weeks. Measurements were collected at baseline and after 12 weeks during the same time of day (±1 hour) in the morning following an overnight fast and abstinence from caffeinated drinks, alcohol, and between 48 and 72 hours after the last exercise session.

ELIGIBILITY:
Inclusion Criteria:

* Stage-1 hypertension
* Postmenopausal

Exclusion Criteria:

* Pulmonary, renal, adrenal, pituitary, severe psychiatric, thyroid, or cardiovascular disease other than stage-1 systolic hypertension (140-159 mmHg)
* Hormone replacement therapy during the 6 months prior the study
* Smoker or having any medication changes in the previous year
* Experience with psychological and physical therapy in the previous year
* History of steady exercise or exercise training in the last year

Ages: 58 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | 12 weeks
  Arterial stiff ness was measured by brachial to ankle pulse wave velocity (baPWV, m/s) using volume plethysmographic device (VP-1000).
Blood pressure (BP) | 12 weeks
  BP (mmHg) was measured by volume plethysmographic device. Diastolic blood pressure and systolic blood pressure were measured.
Muscle strength | 12 weeks
  Muscle strength was measured by the eight repetition maximum (8RM) test using extension machine (Cyber 6000).
Body composition | 12 weeks
  Body composition was measured using eight-polar tactile-electrode impedance meter (InBody 720). Body weight (kg), fat mass (kg), and fat free mass (kg) were assessed.
Height | 12 weeks
  Height (m) was measured with a stadiometer
Heart rate (HR) | 12 weeks
  Heart rate was measured by ECG
Body mass index (BMI) | 12 weeks
  BMI was calculated as weight/height^2 (kg/m^2)

REFERENCES:
- [Derived] Wong A, Figueroa A, Son WM, Chernykh O, Park SY. The effects of stair climbing on arterial stiffness, blood pressure, and leg strength in postmenopausal women with stage 2 hypertension. Menopause. 2018 Jul;25(7):731-737. doi: 10.1097/GME.0000000000001072. PMID 29438269